CLINICAL TRIAL: NCT00808353
Title: Genomic Approaches to Common Chronic Disease
Brief Title: Genomic Approaches to Common Chronic Disease - Ancillary to ARIC
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: University of Texas (Other); Cornell University (Other); Baylor College of Medicine (Other); Washington University School of Medicine (Other)
Responsible Party: Charles F. Sing/Professor, University of Michigan
Other Study IDs: CFDA No: 93.859; 5P50GM065509 (NIH)
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Cardiovascular Disease
Keywords: CVD
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The ARIC study is a prospective epidemiologic study conducted in four U.S. communities and designed to investigate the etiology and natural history of atherosclerosis, the etiology of clinical atherosclerotic diseases, and variation in cardiovascular risk factors, medical care and disease by race, gender, location, and date.

DETAILED DESCRIPTION:
The Atherosclerosis Risk in Communities Study (ARIC), sponsored by the National Heart, Lung and Blood Institute (NHLBI), is a prospective epidemiologic study conducted in four U.S. communities. ARIC is designed to investigate the etiology and natural history of atherosclerosis, the etiology of clinical atherosclerotic diseases, and variation in cardiovascular risk factors, medical care and disease by race, gender, location, and date.

ARIC includes two parts: the Cohort Component and the Community Surveillance Component. The Cohort Component began in 1987, and each ARIC field center randomly selected and recruited a cohort sample of approximately 4,000 individuals aged 45-64 from a defined population in their community. A total of 15,792 participants received an extensive examination, including medical, social, and demographic data. These participants were reexamined every three years with the first screen (baseline) occurring in 1987-89, the second in 1990-92, the third in 1993-95, and the fourth and last exam was in 1996-98. Follow-up occurs yearly by telephone to maintain contact with participants and to assess health status of the cohort.

In the Community Surveillance Component, currently ongoing, these four communities are investigated to determine the community-wide occurrence of hospitalized myocardial infarction and coronary heart disease deaths in men and women aged 35-84 years. Hospitalized stroke is investigated in cohort participants only. The study conducts community surveillance of inpatient heart failure (ages 55 years and older) and cohort surveillance outpatient heart failure events beginning in 2005.

ELIGIBILITY:
Inclusion Criteria:

* The ARIC study began in 1987, and each ARIC field center randomly selected and recruited a cohort sample of approximately 4,000 individuals aged 45-64 from a defined population in their community

Exclusion Criteria:

* Those not meeting the inclusion criteria

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The ARIC study is a prospective epidemiologic study conducted in four U.S. communities The ARIC study began in 1987, with each field center randomly selecting and recruiting a cohort sample of approximately 4,000 individuals aged 45-64 from a defined population in their community. These participants were reexamined every three years with the first screen (baseline) occurring in 1987-89, the second in 1990-92, the third in 1993-95, and the fourth and last exam was in 1996-98. Follow-up occurs yearly by telephone to maintain contact with participants and to assess health status of the cohort.
Sampling Method: Probability Sample
Enrollment: 15792 (Actual)
Dates: Start 1985-07

PRIMARY OUTCOMES:
Cardiovascular disease and its risk factors | One year

SECONDARY OUTCOMES:
Additional common chronic disease risk factors | One year

CONTACTS AND LOCATIONS:
Overall Officials: Eric Boerwinkle, PhD, Principal Investigator — Univeristy of Texas Houston Health Science Center School of Public Health